CLINICAL TRIAL: NCT03939728
Title: Comparison of Lung Ultrasound and Chest Radiography for Pleural and Pulmonary Diagnosis in Pediatric Intensive Care Unit
Acronym: EchoRéaPed
Status: Terminated | Type: Observational
Why Stopped: Investigators on maternity leave and COVID pandemic
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7413
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Pediatric Lung Ultrasound; Pediatric Chest Radiography; Pediatric Lung Diagnosis
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest radiography and lung ultrasound: All patients will be enrolled, during their stay in pediatric intensive care unit, in order to have a pleural or pulmonary diagnosis, a chest radiography and then a lung ultrasound, at less than 2 hours interval.
  Interventions: Radiation: Chest radiography and lung ultrasound

INTERVENTIONS:
Radiation: Chest radiography and lung ultrasound — We'll include all patients which have, during their stay in pediatric intensive care unit, in order to have a pleural or pulmonary diagnosis, a chest radiography and then a lung ultrasound, at less than 2 hours interval.

SUMMARY:
In pediatric intensive care unit of Strasbourg, two exams are easily used for pleural and pulmonary diagnosis : chest radiography, which is the "historic" and reference exam, and commonly systematically the lung ultrasound.

However, chest radiography produces radiation and is less accessible in our unit, because it depends on the radiology department.

On the opposite, the lung ultrasound doesn't produce radiation, is simple, reliable, easily accessible (the investigators have two ultrasound systems in the unit), and simply and quickly achievable at the patient's bedside, including for less experienced operator.

We will evaluate the diagnostic performances of lung ultrasound and chest radiography for pleural and pulmonary diagnosis in pediatric intensive care unit.

ELIGIBILITY:
Inclusion criteria:

* Age under 18 years
* Patient in pediatric intensive care unit
* Patient registered with a social security scheme
* Agreement of the persons entitled to give parental authority over minor
* Patient which has, during his stay in pediatric intensive care unit, in order to have a pleural or pulmonary diagnosis, a chest radiography and then a lung ultrasound, at less than 2 hours interval.

Exclusion criteria:

- Refusal of the patient or of the persons entitled to give parental authority over minor to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient in pediatric intensive care unit, under 18 years old, which has, during his stay, in order to have a pleural or pulmonary diagnosis, a chest radiography and then a lung ultrasound, at less than 2 hours interval.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Kappa-measure | 12 months
  Kappa-measure of concordance between diagnosis obtained by lung ultrasound and chest radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided